CLINICAL TRIAL: NCT02468583
Title: A Double-Blind, Randomized, Parallel Group, Proof of Concept Study Comparing FX006 to Kenalog®-40 in Patients With Post-Traumatic Osteoarthritis of the Knee
Brief Title: Proof of Concept Study Comparing FX006 to Kenalog®-40 in Patients With Post-Traumatic Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2014-007
Record Dates: First submitted 2015-05-27; First posted 2015-06-11 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Post-traumatic Osteoarthritis of the Knee
Keywords: Osteoarthritis; Post-traumatic; Knee; Pain; Corticosteroid; Intra-articular; Injection
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — FX006; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FX006 32mg (Experimental): Single 5 mL intra-articular (IA) injection Extended-release formulation
  Interventions: Drug: FX006 32 mg
- TCA IR 40 mg (Active Comparator): Single 1 mL intra-articular (IA) injection Immediate-release formulation
  Interventions: Drug: TCA IR 40 mg

INTERVENTIONS:
Drug: FX006 32 mg — Experimental
  Other Names: Zilretta
  Arms: FX006 32mg
Drug: TCA IR 40 mg — Comparator
  Other Names: Kenalog®-40; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR 40 mg

SUMMARY:
This study was a double-blind, randomized, parallel group, proof of concept study comparing FX006 to Kenalog®-40 (triamcinolone acetonide injectable suspension, USP) in patients with post-traumatic osteoarthritis of the knee.

DETAILED DESCRIPTION:
This study was a double-blind, randomized, parallel group, proof of concept study patients with post-traumatic osteoarthritis (PTOA) of the knee. Approximately 124 eligible patients were intended to be randomized to one of the two treatment groups (1:1) and treated with a single intra-articular (IA) injection of:

* 32 mg of FX006
* 40 mg of Kenalog®-40 (triamcinolone acetonide injectable suspension, USP)

Each prospective patient underwent a screening evaluation to confirm a diagnosis of PTOA of the knee and concurrence with all other eligibility criteria. Patients were be treated on Day 1 (Baseline) and returned to the clinic at Weeks 4, 8 and 12 for evaluation of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female ≥20 and ≤50 years of age
* Diagnosis of post-traumatic OA of the knee
* Kellgren-Lawrence (K-L) Grade 2 or 3 in the index knee within 6 months prior to or at Screening
* Qualifying mean score on the 24-h average pain score (0-10 numeric rating scale)
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness to abstain from use of restricted medications and therapies during the study

Exclusion Criteria:

* Prior osteotomy of the index knee
* Any condition that could possibly confound the patient's assessment of index knee pain in the judgement of the Investigator (i.e., ipsilateral hip OA, gout, radicular low back pain and hip pain that is referred to the knee that could cause misclassifcation, pain in any other area of the lower extremeties or back that is equal to or greater than the index knee pain)
* Fibromyalgia, Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease
* History of, or clinical signs and symptoms of active infection of the index knee
* Crystal disease of the index knee within one month of Screening
* Disease secondary to surgical treatment of Shatzker grade IV, V, or VI tibial plateau fractures (OTA classification C2 or C3); surgical treatment of OTA calssifcation C2 or C3 distal femur fractures; or >2mm of articular incongruity after surgery
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Intramuscular (IM) or oral corticosteroids (investigational or marketed) within 1 month of Screening
* Any other IA investigational drug/biologic within 6 months of Screening
* Prior use of FX006
* Prior arthroplasty of any type of the index knee or planned/anticipated surgery of the index knee during the study period
* Type 1 or Type 2 diabetes requiring insulin
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, Study Director — Flexion Therapeutics
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FX006 32 mg: 3 subjects received FX006 32 mg as a single 5 mL IA injection
- TCA IR 40 mg: 3 subjects received TCA IR 40 mg as a single 1 mL IA injection
Period: Overall Study
Arm/Group | FX006 32 mg | TCA IR 40 mg
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- FX006 32 mg: FX006: Single 5 mL IA injection
- TCA IR 40 mg: TCA IR: Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 32 mg | TCA IR 40 mg | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 43 [36 to 49] | 40 [37 to 47] | 42 [36 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in the Weekly Mean of the Average Daily (24-hour) Pain Intensity Scores Over Weeks 5 to 10
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine."
Time Frame: 5-10 Weeks
Population: Given that the study was closed early, with only 5% of the planned study population enrolled, efficacy data were not analyzed.
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Weekly Mean of the Average Daily (24-hr) Pain Intensity Scores, Change From Baseline to Each Week and Average Change From Baseline Over Weeks 1 to 12 and Weeks 4 to 12
Description: as for outcome 1
Time Frame: 12 Weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion of Patients Experiencing a >20% Decrease in Pain From Baseline in Weekly Mean of the Average Daily (24-hr) Pain Intensity Scores at Each Week
Time Frame: 12 Weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Patients Experiencing a >50% or >30% Decrease in Pain From Baseline in Weekly Mean of Average Daily 24-hr Pain Intensity Scores at Each Week
Time Frame: 12 Weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion of Patients Experiencing Each of >50% or >30% Decrease in Pain From Baseline in Weekly Mean of the Average Daily (24-hr) Pain Intensity Scores at Each Week
Time Frame: 12 Weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: WOMAC A (Pain Subscale)
Description: change from Baseline to Weeks 4, 8 and 12 average change from Baseline over Weeks 4 to 8 and Weeks 4 to 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: WOMAC A1 (Pain on Walking Question)
Description: change from Baseline to Weeks 4, 8 and 12 average change from Baseline over Weeks 4 to 8 and Weeks 4 to 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: WOMAC B (Stiffness)
Description: change from Baseline to Weeks 4, 8 and 12 average change from Baseline over Weeks 4 to 8 and Weeks 4 to 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: WOMAC C (Function)
Description: change from Baseline to Weeks 4, 8 and 12 average change from Baseline over Weeks 4 to 8 and Weeks 4 to 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: WOMAC (Total):
Description: change from Baseline to Weeks 4, 8 and 12 average change from Baseline over Weeks 4 to 8 and Weeks 4 to 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Knee Injury and Osteoarthritis Score (KOOS)
Description: change from Baseline to Weeks 4, 8 and 12 average change from Baseline over Weeks 4 to 8 and Weeks 4 to 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Patient Global Impression of Change (PGIC) at Weeks 4, 8 and 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Clinical Global Impression of Change (CGIC) at Weeks 4, 8 and 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percent of Responders (Defined as Patients With High Improvement in Pain or Function) According to OMERACT-OARSI Criteria at Weeks 4, 8 and 12
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Time to Onset of Pain Relief
Description: Time to onset of pain relief in days is defined as the time from first dose to the first daily pain assessment showing >30% improvement from the weekly mean of the average daily (24-hr) pain intensity scores at Baseline
Time Frame: Baseline to >30% improvement
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Average Weekly and Total Consumption of Rescue Medication
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | FX006 32 mg | TCA IR 40 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following IA administration through the final study visit at week 12.
Groups:
- TCA IR 40 mg: TCA IR: Single 3 mL IA injection
Arm/Group | FX006 32 mg | TCA IR 40 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 32 mg (N=3) | TCA IR 40 mg (N=3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood triglycerides increased (Infections and infestations) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early with only 5% of the planned study population enrolled, efficacy data were not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes